CLINICAL TRIAL: NCT07363772
Title: Evaluation of Efficacy and Effectiveness of Mixed Reality Cardiopulmonary Resuscitation Training
Brief Title: Evaluation of Mixed Reality Cardiopulmonary Resuscitation Training
Acronym: HEROS 4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ki Jeong Hong, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2401-048-1500
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cardiopulmonary Resuscitation (CPR); Basic Life Support Training Course; Cardiac Arrest (CA)
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEROS 4.0 (Experimental): Participants will receive a two-stage CPR training program consisting of pre-training and on-site MR-based training. As pre-training, participants will be instructed to watch a 40-minute instructional video (conventional CPR training group video) at home prior to their visit. After completing the pre-training, participants will undergo 20 minutes of MR-based CPR training using the HEROS 4.0 system in a dedicated CPR training booth.
  Interventions: Other: HEROS 4.0
- Conventional CPR training (Active Comparator): Participants will receive 60 minutes of standard CPR education delivered through instructional videos and in-person instructor guidance, reflecting current community CPR training practice.
  Interventions: Other: Conventional CPR training

INTERVENTIONS:
Other: HEROS 4.0 — Participants will receive a two-stage CPR training program consisting of pre-training and on-site MR-based training. As pre-training, participants will be instructed to watch a 40-minute instructional video (conventional CPR training group video) at home prior to their visit. After completing the pre-training, participants will undergo 20 minutes of MR-based CPR training using the HEROS 4.0 system in a dedicated CPR training booth. The MR-based CPR training content consists of cardiac arrest recognition, calling emergency medical services, chest compressions, and use of an automated external defibrillator, while minimizing interruptions in chest compressions.
  Arms: HEROS 4.0
Other: Conventional CPR training — Participants will receive 60 minutes of standard CPR education delivered through instructional videos and in-person instructor guidance, reflecting current community CPR training practice.
  Arms: Conventional CPR training

SUMMARY:
<Study Design> This study is a cluster-randomized, stratified, non-inferiority trial designed to evaluate the feasibility, efficacy, and educational effectiveness of HEROS 4.0, a mixed-reality (MR)-based cardiopulmonary resuscitation (CPR) training system, compared with conventional instructor-led CPR training.

<Objective & Hypothesis> The primary objective is to determine whether MR-based HEROS 4.0 CPR training is non-inferior to standard video- and instructor-based CPR training in improving CPR performance quality. The central hypothesis is that participants trained using HEROS 4.0 will achieve comparable CPR quality to those trained using traditional methods, while benefiting from enhanced immersion, scalability, and accessibility.

<Participants> A total of 120 adults aged 18-50 years who have not received CPR training within the previous 12 months will be recruited. Participants will be assigned to one of two clusters and randomized in a 1:1 ratio to either the HEROS 4.0 MR training group or the conventional CPR training group.

<Intervention & Control>

Participants will undergo CPR training according to their assigned group:

Intervention group (HEROS 4.0):

Participants will receive a two-stage CPR training program consisting of pre-training and on-site MR-based training. As pre-training, participants will be instructed to watch a 40-minute instructional video (conventional CPR training group video) at home prior to their visit. After completing the pre-training, participants will undergo 20 minutes of MR-based CPR training using the HEROS 4.0 system in a dedicated CPR training booth.

Control group (Conventional CPR training):

Participants will receive 60 minutes of standard CPR education delivered through instructional videos and in-person instructor guidance, reflecting current community CPR training practice.

<Outcomes> Immediately after training, all participants will undergo a standardized cardiac arrest simulation using a CPR quality-measurement manikin. This simulation will assess objective CPR performance metrics as well as subjective outcomes through questionnaires.

To evaluate knowledge retention and skill durability, all assessments will be repeated 6 months after training using the same simulation scenario and outcome measures.

The primary outcome is chest compression fraction measured during the standardized simulated cardiac arrest scenario.

Secondary outcomes include quantitative measures of CPR quality and participant-reported outcomes based on survey.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years who have not received CPR training within the previous 12 months.

Exclusion Criteria:

* Healthcare professionals
* Individuals unable to safely tolerate MR equipment (e.g. motion sickness)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Chest compression fraction | (1) Immediately after training and (2) at 6-month follow-up.
  Chest compression fraction (CCF) is defined as the proportion of total resuscitation time during which chest compressions are actively delivered. Chest compression quality metrics including CCF will be measured during a standardized cardiac arrest simulation using a CPR quality-measurement manikin.

SECONDARY OUTCOMES:
Mean chest compression depth | (1) Immediately after training and (2) at 6-month follow up.
  The average depth of all chest compressions delivered during the simulated resuscitation.
Mean chest compression rate | (1) Immediately after training and (2) at 6-month follow up.
  The average number of chest compressions performed per minute during the CPR simulation.
Proportion of compressions with adequate depth | (1) Immediately after training and (2) at 6-month follow up.
  The percentage of chest compressions that meet guideline-recommended depth (5-6 cm) criteria during the simulation.
Proportion of compressions with adequate rate | (1) Immediately after training and (2) at 6-month follow up.
  The percentage of chest compressions that fall within the guideline-recommended (100-120 compressions per minute) compression rate range.
Overall basic life support performance | (1) Immediately after training and (2) at 6-month follow up.
  Measurement of basic life support performance during standardized cardiac arrest simulation using the following checklist items including:
  Check response / Assess breathing / Call EMS and get help / Chest compressions / Activate AED and attach pads / Stand clear / Deliver shock / Minimize CPR interruptions /
CPR self-efficacy | (1) Before training, (2) immediately after training and (3) at 6-month follow-up.
  Participants' self-efficacy in performing CPR will be evaluated using a modified version of the Basic Resuscitation Skills Self-Efficacy Scale (BRS-SES), consisting of 15 items rated on a 11-point Likert scale (converted to 0-100 scale), with higher scores indicating greater self-efficacy.
System Usability Scale | Immediately after training
  The usability of the MR-based CPR Training program will be evaluated using the System Usability Scale (SUS), a validated 10-item questionnaire rated on a 5-point Likert scale, with higher scores indicating better usability. This assessment will be conducted only in the experimental group.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Do Shin, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Nowon-gu Public Health Center, Seoul, Nowon-gu, South Korea

IPD SHARING:
Plan to Share IPD: No